CLINICAL TRIAL: NCT03136432
Title: Clinical Determinants of the 6 Minute Walk Test in Children With Cerebral Palsy
Brief Title: Clinical Determinants of the 6 Minute Walk Test in Cerebral Palsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Muserrefe Nur Keles, Research Assistant, Gazi University
Other Study IDs: 8888
Record Dates: First submitted 2017-04-25; First posted 2017-05-02 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Cerebral Palsy; Exercise
Keywords: Cerebral Palsy; Functional Exercise Capacity; Quality of Life
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with cerebral palsy: Children with cerebral palsy, who can walking dependently and continuously for 6 minutes.

SUMMARY:
Cerebral Palsy (CP) is a group of permanent disorders of movement and posture, generally accompanied by secondary musculoskeletal problems. Studies in literature showed taht children with CP supports a link between the levels of impairment and walking ability. The 6 Minute walk test is a standardized, self-placed walking test commonly used to access functional ability in children with cerebral palsy. While decreased exercise capacity has been identified in children with cerebral palsy, the clinical determinants of the 6MWT in this population have not been investigated yet. Thus the aim of this study is to investigate the relationship between 6 Minute walk test, quality of life, respiratory muscle strength,activities of daily living using with Pediatric Evaluation of Disability Inventory and trunk control.

DETAILED DESCRIPTION:
A convenience of children with hemiparetic and diplegia CP, 7-14 years, is going to recruited from Gazi University, Faculty of Health Science, Department of Physiotherapy and Rehabilitation. Every each of patients respiratory muscle strength will be evaluated using with electronic mouth pressure device, trunk control with using trunk control measurement scale, activities of daily living using with Pediatric Evaluation of Disability Inventory (PEDI), functional exercise capacity usin with six minute walk test (6MWT) and quality of life using with Cerebral Palsy Quality of Life Questionnaire (CPQOL).

ELIGIBILITY:
Inclusion Criteria:

* Aged 7-14 years
* Diagnosed to spastic cerebral palsy
* Gross Motor Function Classification System levels I or II.
* Have no earlier interventions in the form of orthopaedic surgery or injection with botulinum toxin type A in the 6 month prior to baseline assessments
* Child are able to demonstrate sufficient co-operation and cognitive understanding participating

Exclusion Criteria:

* Active medical condition impairment (pneumonia etc.)
* Do not accommodate the study
* Do not want to attempt the study

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cerebral palsy who can walk independently continuously for 6 minutes
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2016-12-14 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
Functional exercise capacity | 20 minutes
  6 minute walk test

SECONDARY OUTCOMES:
Respiratory muscle strength | 20 minutes
  Mouth pressure device
Activities of daily living using with Pediatric Evaluation of Disability Inventory | 30 minutes
  PEDI scale
Quality of life | 30 minutes
  CPQOL scale
Change in trunk control over time assessed with Trunk Control Measurement Scale | 20 minutes
  Assessing change in trunk control

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Elbasan, Phd, Study Chair — Gazi University
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University, Faculty of Health and Sciences, Department of Physiotherapy and Rehabilitation Recruiting Ankara, Turkey, 06500, Ankara
  - Gazi University, Faculty of Health and Sciences, Department of Physiotherapy and Rehabilitation, Ankara

IPD SHARING:
Plan to Share IPD: No
we have not decided yet